CLINICAL TRIAL: NCT04545905
Title: Antenatal Care as a Platform for Malaria Surveillance: Utilizing Community Prevalence Measures From the New Nets Project to Validate ANC Surveillance of Malaria in Burkina Faso
Status: Completed | Type: Observational
Sponsor: PATH (Other)
Collaborators: Centre national de recherche et de formation sur le paludisme (Other Government); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 1588786; INV-003761 (Other Grant/Funding Number: Bill & Melinda Gates Foundation)
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-09

CONDITIONS: Malaria
Keywords: Antenatal care; Surveillance; Malaria; Epidemiology; Net use; Net coverage; Prevalence
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women attending first ANC visit: Pregnant women attending their first ANC visit at selected health facilities in Gaoua, Banfora, and Orodara districts.
  Interventions: Diagnostic Test: ANC surveillance

INTERVENTIONS:
Diagnostic Test: ANC surveillance — Clinic-based testing of all pregnant women during antenatal care visits.

SUMMARY:
Burkina Faso will be deploying next-generation ITNs through mass campaigns in pre-determined provinces. As part of New Nets Project's initiative to catalyze the market introduction of next-generation ITNs, enhanced surveillance activities will be conducted to support observational impact analyses. As part of this enhanced surveillance, malaria infection prevalence is being measured through annual cross-sectional surveys during peak transmission periods using rapid diagnostic tests (RDTs) in children aged 6 to 59 months (under 5 years).

It will also include strengthened routine data collection at all health facilities in the districts. The present study aims to leverage the planned cross-sectional surveys and strengthened routine data conducted by the New Nets Project in three of the study districts (Banfora, Gaoua, and Orodara) to assess (1) whether the malaria infection prevalence data collected during antenatal care (ANC) surveillance correlates with these estimates of community infection prevalence in children 6 to 59 months and (2) if intervention coverage data (particularly ITN ownership and use) collected from ANC surveillance are valid and representative of the population as a whole. These additional data could catalyze a new model of surveillance for malaria, and greatly simplify evaluation of the impact of new interventions, as ANC surveillance could potentially replace or supplement cross-sectional household surveys and provide more granular and timely data.

All pregnant women attending first ANC visit at seven health facilities in each study district and who are 20 years old or older or in a union will be eligible for enrollment. Potential participants will be approached during their visit by a health facility worker. During group counselling sessions at initial intake, women will be informed of this pilot surveillance activity, and written informed consent will be obtained from each woman individually prior to routine ANC testing. All consenting women attending ANC first visit at a participating health facilities will be tested for malaria using an RDT and asked to complete a study questionnaire which will include questions about the participant's net use, and care seeking behavior. It is expected to take 15 minutes to complete. Women who test positive for malaria will be given treatment according to national guidelines. There is no additional benefit to individual participants.

The specific objectives of this ANC surveillance pilot are to:

1. Determine the prevalence of malaria infection and coverage of malaria control interventions among pregnant women attending their first ANC visit.
2. Assess the correlation between ANC surveillance parasite prevalence from this study, malaria incidence measured from health facilities, and parasite prevalence collected by the New Nets Project during cross-sectional household surveys.
3. Analyze the correlation between health seeking and net use/access in the ANC surveillance and health seeking behavior compared to the cross-sectional survey

DETAILED DESCRIPTION:
Data from public health surveillance systems are used for multiple purposes, including measuring the burden and monitoring the trends of a disease; guiding the planning, implementation, and evaluation of prevention and control programs; and prioritizing the allocation of health resources. In addition to routine health surveillance activities, public health programs often collect additional data on health indicators , as well as intervention coverage and program utilization, via nationally representative household surveys, such as the Demographic and Health Survey and the Malaria Indicator Survey.

These household surveys provide data to help measure the burden of and monitor trends in malaria, including data on the prevalence of symptomatic and asymptomatic infections in the population. Additionally, because the surveys provide data on monitoring and coverage impact indicators, they help guide the planning, implementation, and evaluation of prevention and control programs, and prioritization of the allocation of national malaria control program (NMCP) resources. Indeed, these representative surveys have become key tools for benchmarking progress towards malaria control and elimination.

Nevertheless, the surveys are expensive to conduct and are limited by long periodic intervals (e.g., every two to five years) and broad sampling strategies (i.e. generating national or regional estimates of disease burden and intervention coverage) that fail to capture seasonal trends or sub-regional heterogeneity, limiting their use for real-time or locally targeted planning and response.

Routine health information systems, on the other hand, may provide a continuous, granular data source representative of all age groups, primarily to help measure the burden and monitor the trends of symptomatic malaria and other diseases. Many countries have implemented standardized, electronic-based health management information system (HMIS), on platforms such as District Health Information System 2, which provide monthly health facility data in real time. Despite being a potential source of valuable public health information, several factors limit the utility of HMIS data and should be considered carefully. One key limitation is the quality and representativity of the data being reported into HMIS, which is affected not only by general data issues, but also by factors such as case management practices and stockouts. These limitations require monitoring and health systems strengthening to overcome. HMIS data on case numbers may also be biased because some symptomatic patients may not present to a facility for care or may not seek care at all, and it can be difficult to interpret the incidence because of uncertainties surrounding regional and local population estimates. Further, not all health facilities report into HMIS; in many countries, the data derive predominantly from public health facilities. If the population using alternative sources of care for diagnosis and treatment of malaria (e.g., private facilities or traditional healers) varies over time, or differs from those using public facilities, the data trends observed in the HMIS may not be representative. Finally, as HMIS data are limited to patients presenting with symptomatic illness, it is not possible to assess the burden and epidemiology of asymptomatic infections, which are believed to represent the majority of malaria infections in many populations. Representativeness and validity of routine data may also be affected by diagnostic testing practices, which in turn may vary by health care provider performance, seasonality, and availability of diagnostic commodities. Finally, data on monitoring and coverage of malaria control interventions, such as insecticide treated bed nets (ITNs), are not typically collected during routine health visits or reported in HMIS.

To build on the strengths and address the limitations of these two complementary surveillance approaches, collecting data on parasite prevalence and coverage of malaria control interventions during antenatal care (ANC) clinic visits may provide an easily accessible, reliable, and representative source for monitoring population trends in malaria control with a higher degree of granularity than is possible in nationally representative household surveys. ANC coverage is high across sub-Saharan Africa; about 90% of women make at least one ANC visit in each pregnancy. Only six countries reported that fewer than 80% of women attended ANC at least once during their most recent pregnancy. Thus, pregnant women attending their first ANC visit are likely to be representative of the overall population of pregnant women. Pregnant women attending their first ANC visit are an ideal population for monitoring trends in malaria prevalence over time, as monthly ANC attendance remains relatively constant over time (minimal effects of seasonality) and is independent of malaria symptoms, thus giving an general infection prevalence estimate similar to that of a community survey. It has been demonstrated that malaria parasite prevalence among pregnant women correlates with the prevalence among children under five years of age. This highlights the possibility that pregnant women could be a good sentinel population for representative measures of trends in malaria prevalence, and raises the question of whether pregnant women would be a good source of data on coverage of malaria control interventions that could be readily tracked over time. Once scaled up, these systems may also provide these data more frequently, at a finer spatial scale, and at a lower cost than household surveys.

In Burkina Faso, the NMCP is distributing new ITNs in mass campaigns in nine provinces. The New Nets Project is funding community surveys in three of these provinces, including rapid diagnostic test (RDT) testing in these provinces, to look at the impact of ITNs. This presents an important opportunity to validate whether the coverage of malaria control interventions and measures of parasite prevalence among pregnant women at first ANC visits is representative of the population at large in Burkina Faso. In three districts, pregnant women presenting for their first ANC visit will be consented and tested for malaria using an RDT and asked to complete a study questionnaire. A comparison of results obtained at first ANC visits will be made to results from concurrent household surveys conducted by the New Nets Project. If validated and found to be a sustainable change to ANC visit procedures, data from the ANC sentinel population could be used to augment or even replace much of the data collected through the use of Malaria Indicator Surveys, which are expensive and infrequently conducted and generally only powered to the regional level. This data could then be triangulated with malaria burden data from the outpatient department to understand variation in community prevalence (as measured through ANC) and malaria clinical incidence, thereby guiding programmatic decision-making and response.

ELIGIBILITY:
Inclusion Criteria:

* Attending ANC first visit at participating health facility
* Pregnant women 20 years or older
* Pregnant women under 20 years old and considered an emancipated

Exclusion Criteria:

• Women with signs of severe malaria as determined by the ANC clinician

Min Age: 20 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Cohorts will be selected from three districts in Burkina Faso: Banfora, Gaoua, Orodara. Malaria is endemic in Burkina Faso, with heightened transmission June and October. The overall malaria incidence per 1,000 people is 722 in Gaoua, 729 in Banfora, and 631 in Orodara. The 2017 Malaria Indicator Survey found that malaria prevalence was 16.9% in children under five, a significant decrease from the 45.7% found during the 2014 survey, though the survey took place after the peak transmission season and could be much higher. Insecticide treated nets are the primary vector control method to prevent malaria and are distributed during mass campaigns, antenatal care and Expanded Programme on Immunizations visits, and in the private sector. Four rounds of seasonal malaria chemoprevention is given to children 3 to 59 months of age between July and October throughout much of the country. An indoor residual spray program was recently restarted 2012 and now covers three high-burden districts.
Sampling Method: Non-Probability Sample
Enrollment: 13350 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
ANC malaria infection prevalence | August 2020 to December 2022
  Malaria infection prevalence among pregnant women attending their first antenatal care visit.

SECONDARY OUTCOMES:
Correlation between cross-sectional and ANC population indicator values | August 2020 to December 2022
  District-level correlation between indicator values estimated from the ANC population and similar estimates from contemporary household cross-sectional surveys conducted by the New Nets Project. These indicators include: RDT confirmed malaria infection prevalence, net access, net use (household), net use (children under 5), prevalence of fever, malaria health care seeking (testing), malaria health care seeking (treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Wagman, PhD, Principal Investigator — PATH
Locations (1):
- Centre National de Recherche et de Formation sur le Paludisme, Ouagadougou, Burkina Faso

REFERENCES:
- [Background] Lindblade KA, Steinhardt L, Samuels A, Kachur SP, Slutsker L. The silent threat: asymptomatic parasitemia and malaria transmission. Expert Rev Anti Infect Ther. 2013 Jun;11(6):623-39. doi: 10.1586/eri.13.45. PMID 23750733
- [Background] van Eijk AM, Hill J, Noor AM, Snow RW, ter Kuile FO. Prevalence of malaria infection in pregnant women compared with children for tracking malaria transmission in sub-Saharan Africa: a systematic review and meta-analysis. Lancet Glob Health. 2015 Oct;3(10):e617-28. doi: 10.1016/S2214-109X(15)00049-2. Epub 2015 Aug 19. PMID 26296450
- [Background] German RR, Lee LM, Horan JM, Milstein RL, Pertowski CA, Waller MN; Guidelines Working Group Centers for Disease Control and Prevention (CDC). Updated guidelines for evaluating public health surveillance systems: recommendations from the Guidelines Working Group. MMWR Recomm Rep. 2001 Jul 27;50(RR-13):1-35; quiz CE1-7. PMID 18634202
- See also: ICF. The DHS Program STATcompiler. Funded by USAID. — http://www.statcompiler.com